CLINICAL TRIAL: NCT05616988
Title: Metabolomic Evaluation of Psycho-surgical Synergy on Body Image Restoration After Breast Cancer
Acronym: BrEva
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Carlo Lai, Full Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URomLS_4
Record Dates: First submitted 2022-10-27; First posted 2022-11-15 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Psychological
Keywords: Mind-Body Intervention; Metabolomics; Breast Reconstruction; Body Image; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will consist of 20 patients with an indication for reconstruction using autologous tissues (DIEP, FALD) and 20 patients with an indication for reconstruction using the immediate prosthesis technique who will carry out the psychological-clinical intervention focusing on expressive writing about their experience of the surgical treatment.
  Interventions: Other: psychological-clinical intervention with three days of expressive writing by Pennebaker
- Control Group (No Intervention): The control group will consist of 20 patients with an indication for reconstruction using autologous tissues (DIEP, FALD) and 20 patients with an indication for reconstruction using the immediate prosthesis technique who will not undergo any kind of psychological-clinical intervention and will be able to apply for the latter at the end of the research.

INTERVENTIONS:
Other: psychological-clinical intervention with three days of expressive writing by Pennebaker — The psychological-clinical intervention involves five interviews with three days of expressive writing by Pennebaker. During the psychological-clinical interviews the following aspects will be explored:
  * Emotions and expectations related to the breast reconstruction process.
  * Feelings related to the perception of one's own body image to promote an integration between the image of one's body and the aspects related to one's own identity and femininity.
  * Thoughts and feelings related to one's relational and social life.
  Expressive writing is a technique devised by Pennebaker (1986), who states that expressing deeper thoughts and feelings through writing can improve the physical and psychological health of the individual. The writing task consists of writing about a traumatic experience or a significant event for the person, for a controlled period (usually 15-30 minutes) and on consecutive days (from 2 to 3 days).
  Arms: Experimental Group

SUMMARY:
The aim of the present study is to verify the effects of a psychological-clinical intervention supported by the technique of expressive writing, on the post-operative course in terms of mental and physical health in patients undergoing surgical mastectomy treatment with post-oncological breast reconstruction. In particular, it is hypothesised that patients undergoing psychological, emotional and social well-being in the phase following surgical treatment, together with an improvement in the inflammatory profile and a possible change in the tryptophan/kynurenine ratio and cortisol.

For this purpose, the recruited patients will be randomly divided into two groups. The first experimental group will consist of 10 patients with an indication for reconstruction using autologous tissues (DIEP, FALD) and 10 patients with an indication for reconstruction using the immediate prosthesis technique who will carry out the psychological-clinical intervention focusing on expressive writing about their experience of the surgical treatment.

The psychological-clinical intervention includes five interviews interspersed with three days of expressive writing by Pennebaker (1986).

The writing task consists of writing about a traumatic experience or an event significant to the person, for a controlled period of time (usually 15 to 30 minutes) and on consecutive days (2 to 3 days).

The second control group will consist of 10 patients with an indication for reconstruction using autologous tissues (DIEP, FALD) and 10 patients with an indication for reconstruction using the immediate prosthesis technique who will not undergo any kind of psychological-clinical intervention and will be able to apply for the latter at the end of the research.

In order to verify the effectiveness of the psychological-clinical intervention, the patients will undergo a psychological evaluation (anxiety, depression, alexithymia, distress, resilience, hope for the future, quality of life, body image, psychological and affective experiences related to breast reconstruction) and a survey of physiological variables (inflammatory response, ratio tryptophan/kynurenine ratio and salivary cortisol) at the various times envisaged in the study: T0 (1 month pre-surgery mastectomy with breast reconstruction), T1(the day after the end of the psychological-clinical intervention), T2 (3 months post psychological-clinical intervention) and T3 (6 months post psychological-clinical intervention).

DETAILED DESCRIPTION:
Breast cancer is the most prevalent cancer globally and is the leading cause of cancer death among women of any age after puberty. Often the diagnosis and treatments of this disease coincide with a long-term worsening of psychophysical well-being, with the following , with consequent impacts on quality-of-life. Among the different treatments, mastectomy with breast reconstruction seems to have relevant effects on psychosocial aspects.

Women with breast cancer show symptoms such as distress, anxiety, depression, and hopelessness for the future, especially between the preliminary diagnosis and the reconstruction surgery.

Furthermore, the psychological and emotional impact concomitant to the treatment pathway can be influenced by the perception of one's body image and aspects related to sexuality.

In cancer patients, this psychological distress can be associated with neurophysiological changes, where an acute state of stress can lead to increased cortisol levels and stimulation of the inflammatory response, thereby increasing the release of numerous pro-inflammatory cytokines and interleukins. All of this may influence the conversion of the essential amino acid tryptophan and its consequent conversion to kynurenine. This psychophysiological interaction appears to play a key role in breast cancer development, progression, metastasis, and therapeutic outcome. Currently, there is evident the need to include a psychological-clinical intervention, supported by the expressive writing technique, within the treatment process for women undergoing surgical mastectomy treatment with breast reconstruction, to bring about an increase in patients' awareness and efficiency and improve their general health status. Moreover, the psychological-clinical intervention could modulate the complex metabolic and inflammatory responses of the body that characterize the oncological condition, going to improve psychophysical well-being.

The main objective of this study is to verify the effects of a psychological-clinical intervention supported by the expressive writing technique, on the post-operative course in terms of mental and physical health in patients undergoing post-oncological breast reconstruction. In particular, the present study intends to combine the evaluation of the therapeutic process through specific psychological scales with the variations of the phenotypic profile, based on the evaluation by Point Of Care Testing (POCT) of physiological parameters of interest, such as the values of inflammatory markers (Serum Amyloid A and IL-6), the tryptophan/kynurenine ratio and cortisol levels. It is hypothesised that patients undergoing the psychological-clinical intervention improve their psychological, emotional, and social well-being in the phase following the surgical treatment, together with an improvement in the inflammatory profile and a possible change in the tryptophan/kynurenine ratio and cortisol.

This study and its results will prompt an innovative multidisciplinary view of the psychophysical well-being of the woman involved in the post-oncological reconstructive care path. Patients' health will be pursued through the integration of the reconstructed part of the breast which will be evaluated on a phenotypic level, general aspects taking into account both psychological and biological ones.

80 female patients undergoing mastectomy surgery with post-oncological breast reconstruction will be recruited at the Plastic Surgery Unit (OU) of the Sant'Andrea Hospital, Faculty of Medicine and Psychology "La Sapienza'' University of Rome. Patients will be required to participate voluntarily, free of charge and informed consent will be required.

During the first consultation, the indication for the type of reconstruction (autologous vs immediate prosthesis) will be decided on the basis of the type of mastectomy and the characteristics of the patient.

Depending on the type of reconstruction, patients will be randomly assigned to the following groups:

* Experimental Group A: 20 patients with indications for reconstruction using autologous tissues (DIEP, FALD) who will carry out the psychological-clinical intervention focused on expressive writing about their experience of surgical treatment.
* Control Group B: 20 patients with indication for reconstruction using autologous tissues (DIEP, FALD) who will not perform any psychological-clinical intervention.
* Experimental Group C: 20 patients with an indication for reconstruction using the direct to implant reconstruction who will carry out the psychological-clinical intervention focused on expressive writing about their experience of surgical treatment.
* Control Group D: 20 patients with indication for reconstruction using the direct to implant reconstruction who will not perform any psychological-clinical intervention.

Patients in the control group will be able to apply for the psychological-clinical intervention at the end of the research.

In the first phase of the study, patients meeting the inclusion criteria will be identified and ask them to sign informed consent for participation in the study. All patients included in the study will undergo a preliminary visit before surgery where they will receive standardised laboratory and radiologic exams needed to establish eligibility for surgery.

Furthermore, will carry out a first measurement of the variables of interest of the study. Measurements will include a salivary matrix sample, a blood sample and the battery of psychological questionnaires.

Subsequently, all patients will be admitted to the department of Plastic Surgery the day before surgery, and they will be asked to sign the informed consent for surgery and then preoperative markings will be performed by the surgeon. The patients will be discharged based on the type of reconstruction and the postoperative status between the 1st and 3rd postoperative day. Finally, the patients will be randomized to double-blind research groups (experimental and control).

In the second phase of the study, corresponding to the post-operative period, the experimental group is scheduled for five weekly interviews interspersed with three days of expressive writing by Pennebaker (1986).

Following the first three psychological-clinical interviews, the three days of expressive writing will be carried out. During these days the patients of the experimental group will be asked to write, for 20 minutes a day, their deepest emotions, thoughts, and concerns related to the surgical treatment.

The patients of the experimental group will carry out the expressive writing session in their homes, in a closed, silent room, which guarantees their privacy.

In the last two psychological-clinical interviews, the emotional aspects that emerged during the three days of expressive writing will also be discussed with the patient.

No psychological-clinical intervention is envisaged for the control group, which can be requested at the end of the research.

In addition, the concentrations of the different metabolites of the kynurenine pathway involved in inflammatory processes and concomitant psychopathological mechanisms. In particular, the dosages will be carried out on a salivary matrix collected immediately before and 30 minutes after the psychological-clinical session. The results will be normalized through the acquisition of the values of inflammation markers such as SAA and IL-6.

The day after the end of the psychological-clinical intervention (T1) and in the various follow-up months (T2, T3), a salivary sample and a capillary blood sample will be taken from each patient, and will also be asked to fill out again the battery of questionnaires previously reported.

ELIGIBILITY:
Inclusion Criteria:

* Presence of diagnosis of breast cancer
* indication to undergo surgical mastectomy treatment
* Italian nationality
* level of education not lower than a secondary school diploma, ensuring sufficient writing skills.

Exclusion Criteria:

* the occurrence of metastases and/or relapse during the study phase,
* the refusal of patients to undergo reconstruction treatment
* the presence of existing psychopathological diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change of Depressive symptoms | 6 months
  In order to test any variation in depressive symptoms the Beck Inventory Scale - BDI was administered in the pre-operative phase (T0), on the day after the end of the clinical psychological intervention (T1) and at the 3-month (T2) and 6-month follow-ups (T3). The Scores 0-13 indicate an absence of depressive content, the scores between 14-19 a mild depression, the scores 27-29 a moderate grade depression and the scores 30-63: a severe depression.
  We will expect a lower level of depression in those who carried out clinical psychology intervention with expressive writing task.
Change of Anxiety Levels | 6 months
  In order to test any variation in anxiety levels all participants completed State-Trait Anxiety Inventory - STAI in the pre-operative phase (T0), on the day after the end of the clinical psychological intervention (T1) and at the 3-month (T2) and 6-month follow-ups (T3). The scores between 80-71 represent very high level of state and trait anxiety, 70-51 represent medium-high level, 50-31 represent medium-low level and 30-20 none or very low level.
  We expected lower level of anxiety in those who carried out clinical psychology intervention with expressive writing task.
Change of Alexithymia | 6 months
  In order to evaluate the level of alexithymia the TAS-20 will be administered in the pre-operative phase (T0), on the day after the end of the clinical psychological intervention (T1) and at the 3-month (T2) and 6-month follow-ups (T3). It is a self-administered questionnaire, consisting of 20 items. The scale ranges between 20 to 100 and it allows to identify alexithymic (> 60), not alexithymic (< 51) and probably alexithymic patients (51-60).
  We will expect lower level of difficulties in identifying, recognizing and describing emotions in those who carried out clinical psychology intervention with expressive writing task.
Change of Resilience | 6 months
  In order to investigate resilience, all participants completed 14-item Resilience Scale - RS-14 in the pre-operative phase (T0), on the day after the end of the clinical psychological intervention (T1) and at the 3-month (T2) and 6-month follow-ups (T3). Higher scores mean superior levels of resilience tendencies.
  We will expect higher level of resilience in those who carried out clinical psychology intervention with expressive writing task.
Change of Psychological distress | 6 months
  In order to investigate the impact of oncological disease and treatment in terms of psychological distress, all participants completed Psychological Distress Inventory - PDI in the pre-operative phase (T0), on the day after the end of the clinical psychological intervention (T1) and at the 3-month (T2) and 6-month follow-ups (T3). High scores correspond to a high degree of distress perceived by the subject.
  We will expect lower level of distress in those who carried out clinical psychology intervention with expressive writing task.
Change of People's Dispositional Optimism | 6 months
  In order to investigate how optimistic or pessimistic people feel about the future, all participants completed Life Orientation Test Revised - LOT-R in the pre-operative phase (T0), on the day after the end of the clinical psychological intervention (T1) and at the 3-month (T2) and 6-month follow-ups (T3). Scores range from zero to 24; higher scores indicate greater optimism and lower scores indicate lower optimism, often referred to as pessimism.
  We will expect higher level of optimism in those who carried out clinical psychology intervention with expressive writing task.
Change of Hopelessness | 6 months
  In order to investigate hope for the future in the participants, the Beck Hopelessness Scale - BHS will be administered in the pre-operative phase (T0), on the day after the end of the clinical psychological intervention (T1) and at the 3-month (T2) and 6-month follow-ups (T3). Higher scores indicate the increased respondent's negative expectations for the future.
  We will expect lower level of negative attitudes, or pessimism, about the future in those who carried out clinical psychology intervention with expressive writing task.
Change of Body Image | 6 months
  In order to investigate the discomfort related to the one's body image, all participants completed Body Uneasiness Test - BUT in the pre-operative phase (T0), on the day after the end of the clinical psychological intervention (T1) and at the 3-month (T2) and 6-month follow-ups (T3). Higher ratings indicate higher levels of body uneasiness.
  We will expect lower level of body uneasiness in those who carried out clinical psychology intervention with expressive writing task.
Change of Breast Cancer Core | 6 months
  In order to investigate expectations, results and experience of women undergoing breast cancer surgery, all participants completed BREAST-Q in the pre-operative phase (T0), on the day after the end of the clinical psychological intervention (T1) and at the 3-month (T2) and 6-month follow-ups (T3).
  We will expect greater satisfaction and better health-related quality of life in those who carried out clinical psychology intervention with expressive writing task.

SECONDARY OUTCOMES:
Change of kynurenine/tryptophan ratio | 6 months
  Physiological parameters related to the kynurenine/tryptophan ratio will be determined in a salivary matrix and assessed by POCT.
Change of Cortisol | 6 months
  Physiological parameters related to the cortisol will be determined in a salivary matrix and assessed by POCT.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lai, Principal Investigator — Department of Dynamic and Clinical Psychology, and Health Studies Sapienza University of Rome
Locations (1):
- Sant'Andrea Hospital, Faculty of Medicine and Psychology "La Sapienza'' University of Rome, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data was collected and stored by the Dynamics department and clinical psychology laptop, protected by a password. The data are accessible only to the Chief Researcher, the Ph.D. student, and the secondary researcher.
  The study protocol will be shared with other sub-investigators involved in the study, but not sensitive data. The study report will be shared and published in a scientific journal, but the privacy of each participant will be respected according to the agreements established by the ethics committee.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 24 months
Access Criteria: The sensitive data are collected in an excel database on the department of Dynamic and Clinical psychology laptop, protected by a password. Each participant is identified by a personal numerical code, to guarantee them their privacy. All the sensitive data will be accessible only by the Chief investigator, the Ph.D. student, and the sub-investigator co-responsible for the study.